CLINICAL TRIAL: NCT00372541
Title: Ceftriaxone Versus Chloramphenicol for Treatment of Severe Pneumonia in Children Aged Less Than Five Years at Mulago Hospital: A Randomized Controlled Trial
Brief Title: Ceftriaxone Versus Chloramphenicol for Treatment of Severe Pneumonia in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Makerere University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HD1120041348U
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2010-07

CONDITIONS: Pneumonia
Keywords: ceftriaxone; chloramphenicol; severe pneumonia; children
MeSH Terms: conditions — Pneumonia | interventions — Ceftriaxone

INTERVENTIONS:
Drug: ceftriaxone

SUMMARY:
Acute lower respiratory tract infections are a leading cause of morbidity and mortality in sub Saharan Africa. The World Health Organisation (WHO) still recommends intravenous chloramphenicol for the treatment of severe pneumonia in children aged less than five years. However, up to 20% of children fail treatment due to the emergence of resistance by bacteria. Several centers now use ceftriaxone, a third generation cephalosporin, which is reported to be efficacious in the treatment of severe pneumonia. However the high cost of ceftriaxone is too prohibitive to allow for its routine use in resource constrained countries. The purpose of this study is to compare chloramphenicol and ceftriaxone in the treatment of severe pneumonia in children under five.

We hypothesize that 92.7% of children who receive once daily intravenous ceftriaxone (75 mg/kg body weight)for 7 days, will recover from severe pneumonia compared to 80.2 % of those who receive intravenous chloramphenicol (25mg/kg body weight/dose every 6 hours for 7 days).

DETAILED DESCRIPTION:
A recent report from the World health Organization showed pneumonia was the leading cause of death in children less than 5 years. WHO recommends intravenous Chloramphenicol 25mg/kg six hourly as the first line drug for the treatment of severe pneumonia in these children. Ceftriaxone 75mg/kg daily is the second line drug.

The efficacy of chloramphenicol for the treatment of severe pneumonia ranges from 80%-84%, while that of ceftriaxone ranges from 85% to 97%. However the high cost of ceftriaxone is too prohibitive to allow for its routine use in resource constrained countries. A study comparing penicillin G plus chloramphenicol and ceftriaxone in the treatment of severe pneumonia in Turkey found that both drugs were equally effective in normalization of the outcome parameters. A recent Cochrane review found no randomized controlled trials comparing both drugs in the treatment of severe forms of pneumonia.

The objective of this study it to compare the efficacy of Ceftriaxone versus Chloramphenicol in the treatment of severe pneumonia in the children under five years of age admitted to Mulago hospital.

This will be a double- blinded randomized controlled trial. Three hundred forty eight children with severe pneumonia will be randomized to receive either intravenous ceftriaxone 75mg/kg/day for seven days or intravenous chloramphenicol 100mg/kg/day for seven days. The primary outcome will mortality and secondary outcomes will be time taken to normalization of respiratory rate, temperature and oxygen saturation.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 months to 59months with cough, difficult breathing and lower chest indrawing
* Consent from parent/carer

Exclusion Criteria:

* Children with severe Asthmatic attack
* Allergy to any of the study drugs
* Diagnosis of Pneumocystis JiroveciPneumonia on therapeutic treatment

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 348 (Estimated)
Dates: Start 2006-09; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Mortality from severe pneumonia by 7th day of treatment

SECONDARY OUTCOMES:
Time to normalisation of respiratory rate
Time to normalisation temperature
Time to normalisation of oxygen saturation

CONTACTS AND LOCATIONS:
Overall Officials: Cordelia M Katureebe, MBCHB, Principal Investigator — Makerere University
Locations (4):
- Uganda (4):
  - Department of Paediatrics and Child Health, Mulago Hospital, Kampala, East Africa
  - Department of Paediatrics and Child Health, Makerere University, Kampala, Kampala
  - Department of paediatrics and child Health,Makerere university, Kampala, Kampala
  - Department of Paediatrics and Child, Makerere University, Kampala, Kampala

REFERENCES:
- [Background] Cetinkaya F, Gogremis A, Kutluk G. Comparison of two antibiotic regimens in the empirical treatment of severe childhood pneumonia. Indian J Pediatr. 2004 Nov;71(11):969-72. doi: 10.1007/BF02828108. PMID 15572814
- [Background] Bakeera-Kitaka S, Musoke P, Downing R, Tumwine JK. Pneumocystis carinii in children with severe pneumonia at Mulago Hospital, Uganda. Ann Trop Paediatr. 2004 Sep;24(3):227-35. doi: 10.1179/027249304225019046. PMID 15479572
- [Background] Bjerre LM, Verheij TJ, Kochen MM. Antibiotics for community acquired pneumonia in adult outpatients. Cochrane Database Syst Rev. 2004;(2):CD002109. doi: 10.1002/14651858.CD002109.pub2. PMID 15106168
- [Background] Ortiz-Ruiz G, Vetter N, Isaacs R, Carides A, Woods GL, Friedland I. Ertapenem versus ceftriaxone for the treatment of community-acquired pneumonia in adults: combined analysis of two multicentre randomized, double-blind studies. J Antimicrob Chemother. 2004 Jun;53 Suppl 2:ii59-66. doi: 10.1093/jac/dkh207. PMID 15150184